CLINICAL TRIAL: NCT07365098
Title: Assessment of Functional Capacity in Liver Transplant Recipients Using the 30-Second Lie-to-Sit Test
Brief Title: Liver Transplant Recipients and 30-Second Lie-to-Sit Test
Status: Recruiting | Type: Observational
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, BÜŞRA CANDİRİ, Assistant Professor, Inonu University
Other Study IDs: 2025/8550
Record Dates: First submitted 2026-01-15; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-11

CONDITIONS: Liver Transplant Recipients
Keywords: liver; functional capacity; liver transplant recipients; 30 second lie-to-sit test
MeSH Terms: interventions — Waist Circumference

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: 30-second lie-to-sit test — In this test, participants will be asked to start from a supine position with their head and arms supported and move to a sitting position as quickly as possible.
  They will be allowed to use one hand and, if necessary, a thin cushion to help them sit up. The number of repetitions performed within 30 seconds will be recorded.
Other: Modified Borg Scale — Following the 30-second lie-to-sit test, the modified Borg scale will be used to assess participants' perceived exertion levels.This scale is a standard tool that allows individuals to subjectively assess their level of exertion during physical activity or exercise, rated from 0 (no exertion) to 10 (maximum exertion).
Other: waist circumference — Waist circumference will be measured in centimeters at the narrowest point between the lowest rib and the upper border of the pelvis while the participant is standing, and the value will be recorded.
Other: 30-second sit-to-stand test — The 30-second sit-to-stand test will be used to assess participants' lower extremity muscle strength and functional capacity. In this test, the participant sits with their back against a chair, feet flat on the floor, and arms crossed over the chest, and stands up and sits down as many times as possible within 30 seconds. Hands should not touch the chair during the test, and only full, complete repetitions are counted. The total number of repetitions at the end of the test will be recorded.
Other: Quadriceps muscle strength — Quadriceps muscle strength will be measured isometrically using a hand-held dynamometer. The participant will be seated with the knees flexed at 90°. The dynamometer will be placed on the front of the leg at ankle level, and the participant will be asked to lift the leg with maximal effort. Three measurements will be taken for each leg, and the average value will be recorded.
Other: Deltoid muscle strength — Isometric strength of the deltoid muscle will be assessed using a hand-held dynamometer. The participant will be seated with the shoulder positioned at 90° abduction and the elbow slightly flexed. The dynamometer will be placed on the lateral side of the upper arm at elbow level, and the participant will perform maximum-effort shoulder abduction. Three measurements will be taken for each extremity, and the average value will be recorded.
Other: Trunk flexion strength — The isometric trunk flexion strength test will be performed with the participant positioned supine, with the knees extented or the hips flexed at 30°. The dynamometer will be placed below the suprasternal notch of the sternum. The participant will place their hands on the opposite acromions and perform isometric trunk flexion.
Other: Trunk extension strength — The isometric trunk extension strength, the participant will be positioned prone while lying down. The dynamometer will be placed at the T4 level, and the participant will be asked to perform maximum isometric trunk extension. In each test position, participants will first perform a submaximal trial, followed by three correct repetitions, and the average value will be recorded.
Other: Handgrip strength — Handgrip strength will be assessed using a hand dynamometer. Participants will be seated with their shoulders adducted at the sides, elbows flexed at 90°, forearms in a neutral position, and wrists positioned at 0-30° extension and 0-15° ulnar deviation. Three trials will be performed for each hand, with a 30-second rest between trials. For analysis, the average of three measurements for both hands will be recorded.
Other: 2-minute walk test — The 2-minute walk test will be used to assess participants' exercise capacity and physical performance. During the test, participants will walk at a self-selected, safe pace for two minutes, and the distance covered in meters will be recorded.
Other: Upper Extremity Functional Index-15 (UEFI-15) — This questionnaire consists of 15 items that assess difficulties in using the upper extremities for activities of daily living. Each item is scored from 0 (cannot do) to 4 (no difficulty). The raw score ranges from 0 to 59 and is converted to a final score ranging from 0 to 100. A higher final score indicates better upper extremity function, providing a comprehensive assessment of functional capacity.
Other: Lower Extremity Functional Scale (LEFS) — This questionnaire is important for assessing lower extremity functional capacity and examining activity limitations in various lower extremity disorders. It consists of 20 items, each scored from 0 (extreme difficulty or unable to perform the activity) to 4 (no difficulty). Intermediate values are defined as 1 (quite difficult), 2 (moderately difficult), and 3 (somewhat difficult). The total score ranges from 0 to 80, with higher scores indicating better functional level.

SUMMARY:
The aim of this study is to assess functional capacity in liver transplant recipients using the 30-second lie-to-sit test and to examine the relationships between functional capacity and variables such as muscle strength, upper and lower extremity function, exercise capacity, and perceived exertion.

DETAILED DESCRIPTION:
Participants' demographic and clinical characteristics, including age, gender, BMI, waist circumference, and relevant clinical data, will be recorded. Functional capacity will also be assessed using the 30-second sit-to-stand test, the 2-minute walk test, and upper and lower extremity functional scales (UEFI-15, AEFÖ), with perceived exertion measured using the Modified Borg Scale. Muscle strength will be measured isometrically with a dynamometer for the quadriceps, deltoid, trunk flexor/extensor muscles, and handgrip. The obtained data will provide a comprehensive evaluation of muscle strength and functional status, contributing to individualized rehabilitation planning.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years
* Diagnosed with end-stage liver disease and listed for liver transplantation
* Ability to speak, understand, and write in Turkish
* No mental disorders
* Voluntary participation with informed consent

Exclusion Criteria:

* Pulmonary, neurological, or cardiac diseases that may interfere with adherence to the assessment protocol
* Difficulty complying with the assessment program
* Musculoskeletal problems
* History of regular physical activity
* Multiple organ failure
* Cognitive impairment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: liver transplant recipients
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2025-11-08 (Actual); Primary Completion 2026-10-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
30-second lie-to-sit test | 24 hours
  In this test, participants will be asked to start from a supine position with their head and arms supported and move to a sitting position as quickly as possible. They will be allowed to use one hand and, if necessary, a thin cushion to help them sit up. The number of repetitions performed within 30 seconds will be recorded.

SECONDARY OUTCOMES:
Waist Circumference | 24 hours
  Waist circumference will be measured in centimeters at the narrowest point between the lowest rib and the upper border of the pelvis while the participant is standing, and the value will be recorded.
Modified Borg Scale | 24 hours
  Following the 30-second lie-to-sit test, the modified Borg scale will be used to assess participants' perceived exertion levels.This scale is a standard tool that allows individuals to subjectively assess their level of exertion during physical activity or exercise, rated from 0 (no exertion) to 10 (maximum exertion).
30-second sit-to-stand test | 24 hours
  The 30-second sit-to-stand test will be used to assess participants' lower extremity muscle strength and functional capacity. In this test, the participant sits with their back against a chair, feet flat on the floor, and arms crossed over the chest, and stands up and sits down as many times as possible within 30 seconds. Hands should not touch the chair during the test, and only full, complete repetitions are counted. The total number of repetitions at the end of the test will be recorded.
Quadriceps muscle strength | 24 hours
  Quadriceps muscle strength will be measured isometrically using a hand-held dynamometer. The participant will be seated with the knees flexed at 90°. The dynamometer will be placed on the front of the leg at ankle level, and the participant will be asked to lift the leg with maximal effort. Three measurements will be taken for each leg, and the average value will be recorded.
Deltoid muscle strength | 24 hours
  Isometric strength of the deltoid muscle will be assessed using a hand-held dynamometer. The participant will be seated with the shoulder positioned at 90° abduction and the elbow slightly flexed. The dynamometer will be placed on the lateral side of the upper arm at elbow level, and the participant will perform maximum-effort shoulder abduction. Three measurements will be taken for each extremity, and the average value will be recorded.
Trunk flexion strength | 24 hours
  The isometric trunk flexion strength test will be performed with the participant positioned supine, with the knees extented or the hips flexed at 30°. The dynamometer will be placed below the suprasternal notch of the sternum. The participant will place their hands on the opposite acromions and perform isometric trunk flexion.
Trunk extension strength | 24 hours
  The isometric trunk extension strength, the participant will be positioned prone while lying down. The dynamometer will be placed at the T4 level, and the participant will be asked to perform maximum isometric trunk extension. In each test position, participants will first perform a submaximal trial, followed by three correct repetitions, and the average value will be recorded.
Handgrip strength | 24 hours
  Handgrip strength will be assessed using a hand dynamometer. Participants will be seated with their shoulders adducted at the sides, elbows flexed at 90°, forearms in a neutral position, and wrists positioned at 0-30° extension and 0-15° ulnar deviation. Three trials will be performed for each hand, with a 30-second rest between trials. For analysis, the average of three measurements for both hands will be recorded.
2-minute Walk Test | 24 hours
  The 2-minute walk test will be used to assess participants' exercise capacity and physical performance. During the test, participants will walk at a self-selected, safe pace for two minutes, and the distance covered in meters will be recorded.
Upper Extremity Functional Index-15 (UEFI-15) | 24 hours
  This questionnaire consists of 15 items that assess difficulties in using the upper extremities for activities of daily living. Each item is scored from 0 (cannot do) to 4 (no difficulty). The raw score ranges from 0 to 59 and is converted to a final score ranging from 0 to 100. A higher final score indicates better upper extremity function, providing a comprehensive assessment of functional capacity.
Lower Extremity Functional Scale (LEFS) | 24 hours
  This questionnaire is important for assessing lower extremity functional capacity and examining activity limitations in various lower extremity disorders. It consists of 20 items, each scored from 0 (extreme difficulty or unable to perform the activity) to 4 (no difficulty). Intermediate values are defined as 1 (quite difficult), 2 (moderately difficult), and 3 (somewhat difficult). The total score ranges from 0 to 80, with higher scores indicating better functional level.

CONTACTS AND LOCATIONS:
Locations (1):
- Inonu Unıversity, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No